CLINICAL TRIAL: NCT02180451
Title: Observational Study to Investigate the Melatonin and Cortisol Circadian Rhythms of Individuals With Smith-Magenis Syndrome (SMS)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: VP-1401
Record Dates: First submitted 2014-06-09; First posted 2014-07-02 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Smith Magenis Syndrome
MeSH Terms: conditions — Smith-Magenis Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Melatonin and Cortisol samples will be collected
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to characterize the circadian rhythm disruption experienced by patients as determined by plasma melatonin, cortisol, and other circadian analytes

ELIGIBILITY:
Inclusion Criteria:

* A confirmed clinical diagnosis of SMS with a prior positive genetic test result as indicated by a parent/guardian
* Informed consent from the patient or the legal guardian/assent provided by the individual with SMS, when possible
* Male or female between the ages of 6-50 years of age
* History of sleep disturbances
* Willing and able to comply with study requirements and restrictions

Exclusion Criteria:

* Failure to confirm diagnosis of SMS by molecular cytogenetic methods and/or DNA-based mutation analysis of the RAI1 gene
* Totally blind with no light perception
* Institutionalized or living in an assisted living facility
* Unwilling or unable to follow medication restrictions (medications that affect sleep or melatonin secretion) or unwilling or unable to sufficiently wash-out from use of a restricted medication
* Any medical condition, as determined by the clinical investigator that would make it unsafe for blood draws (e.g., anemia, blood clotting disorders, anxiety, etc.)
* Any other sound medical reason as determined by the clinical investigator

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Smith-Magenis patients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-06; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Circadian melatonin rhythm as measured by plasma melatonin | 36-hour blood sampling on week 1
Circadian melatonin rhythm as measured by plasma melatonin | 36-hour blood sampling on week 2
Circadian melatonin rhythm as measured by plasma melatonin | 36-hour blood sampling on week 4
Circadian cortisol rhythms as measured by plasma cortisol | 36-hour blood sampling at week 1
Circadian cortisol rhythms as measured by plasma cortisol | 36-hour blood sampling at week 2
Circadian cortisol rhythms as measured by plasma cortisol | 36-hour blood sampling at week 4
Circadian analytes rhythms as measured in plasma | 36-hour blood sampling at week 1
Circadian analytes rhythms as measured in plasma | 36-hour blood sampling at week 2
Circadian analytes rhythms as measured in plasma | 36-hour blood sampling at week 4

SECONDARY OUTCOMES:
Genetic testing to confirm SMS diagnosis | blood sampling at screening visit
Nighttime and daytime sleep as measured by actigraphy | Four week evaluation period
QOL Scale | Four week evaluation period
Melatonin Light Response Test (MLRT) | After four week evaluation period
Behavioral Scale | Four week evaluation period
Salivary melatonin and cortisol | Four week evaluation period

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore, Maryland, United States